CLINICAL TRIAL: NCT03591133
Title: Phase I Clinical Study of TS-143 in Healthy Adult Male Subjects (Single-Dose Administration)
Brief Title: Clinical Study of TS-143 in Healthy Adult Male Subjects (Single-Dose Administration)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TS143-01-01
Record Dates: First submitted 2018-04-18; First posted 2018-07-19 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-06

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Step1:3㎎ QD (Other): Drug: TS-143 3mg Drug: Placebo
  Interventions: Drug: TS-143; Drug: Placebo
- Step2:6㎎ QD (Other): Drug: TS-143 6mg Drug: Placebo
  Interventions: Drug: TS-143; Drug: Placebo
- Step3-1:11㎎ QD (Other): Drug: TS-143 11mg Drug: Placebo
  Interventions: Drug: TS-143; Drug: Placebo
- Step3-2:11㎎ QD（Fed) (Other): Drug: TS-143 11mg Drug: Placebo
  Interventions: Drug: TS-143; Drug: Placebo
- Step4:20㎎ QD (Other): Drug: TS-143 20mg Drug: Placebo
  Interventions: Drug: TS-143; Drug: Placebo
- Step5:36㎎ QD (Other): Drug: TS-143 36mg Drug: Placebo
  Interventions: Drug: TS-143; Drug: Placebo

INTERVENTIONS:
Drug: TS-143
Drug: Placebo

SUMMARY:
To investigate the safety, pharmacokinetics and pharmacodynamics when administering a single dose of TS-143 to Japanese healthy adult males using a placebo-controlled, double-blind, dose-ascending study, in addition to the effects of meals.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with a body-mass index (BMI) of 18.5 to less than 25.0 at the time of the screening tests
2. Subjects judged by the principal investigator or a subinvestigator to be appropriate for participation in the study based on the results of the screening tests and the tests conducted prior to the investigational drug treatment

Exclusion Criteria:

1. Subjects who meet any of the following criteria in the screening tests or the tests conducted on Day -1 and prior to the investigational drug treatment

   * Red blood cell count: ≥ 535 × 10^4 /μL
   * Hemoglobin: ≥ 16.2 g/dL
   * Hematocrit: ≥ 47.5%
   * Reticulocyte ratio: Outside of the reference value range
2. Subjects who meet any of the following criteria in the screening tests

   * Serum EPO concentration: Outside of the reference value range
   * Ferritin: 30 ng/mL or less, or ≥ 262 ng/mL
3. Subjects who meet any of the following criteria in the vital signs in the screening tests and the tests conducted prior to the investigational drug treatment

   * Blood pressure: Systolic blood pressure ≥ 140 mmHg, or diastolic blood pressure ≥ 90 mmHg or more
   * Pulse rate: < 40 bpm, or ≥ 100 bpm
   * Body temperature: ≥ 37.5°C

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-24 (Actual); Primary Completion 2016-04-14 (Actual); Study Completion 2016-04-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 8 days
  To evaluate the safety of TS-143 given single administration in healthy volunteers by incidence of adverse events which include abnormal electrocardiograms, vital signs, and clinical laboratory parameters.
Plasma concentrations of unchanged form (ng/mL) | 72 hours
  The descriptive statistics (e.g., number of subjects, arithmetic mean, standard deviation) were calculated by dose group and evaluation timing.
Urinary excretions of unchanged form (ng/mL) | 72 hours
  The descriptive statistics (e.g., number of subjects, arithmetic mean, standard deviation) for the total urinary excretion (amount and fraction) were summarized by dose group.
Serum erythropoietin (EPO) concentration | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Okuyama, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shinfuku A, Shimazaki T, Fujiwara M, Sato F, Watase H, Numazaki T, Kawakita Y, Mutoh M, Yamasaki H, Takayama N, Kato S, Sugimoto T, Maruyama J. Novel Compound Induces Erythropoietin Secretion through Liver Effects in Chronic Kidney Disease Patients and Healthy Volunteers. Am J Nephrol. 2018;48(3):157-164. doi: 10.1159/000492181. Epub 2018 Sep 3. PMID 30176654